CLINICAL TRIAL: NCT04561375
Title: A Pilot Study Assessing the Effects of Sublingual Sufentanil 30 µg on Postoperative Recovery From Ambulatory Surgery
Brief Title: Assessing the Effects of Sublingual Sufentanil 30 µg on Postoperative Recovery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: For practical reasons of slow enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-642
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthroscopy
MeSH Terms: interventions — Sufentanil; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): 30 µg tablet of sublingual sufentanil preoperatively and fentanyl placebo at induction of anesthesia.
  Interventions: Drug: Sufentanil
- Control Group (Placebo Comparator): placebo sublingual sufentanil preoperatively and 50 µg fentanyl at induction of anesthesia
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Sufentanil — 30 µg tablet of sublingual sufentanil
  Arms: Intervention Group
Drug: Fentanyl — 50 µg fentanyl
  Arms: Control Group

SUMMARY:
A pilot study to evaluate the effect of incorporating sublingual sufentanil into our perioperative opioid regimen for ambulatory orthopedic surgery.

DETAILED DESCRIPTION:
A pilot study to evaluate the effect of incorporating sublingual sufentanil into our perioperative opioid regimen for ambulatory orthopedic surgery. The results will help us estimate treatment effect and determine sample size for a subsequent full-scale clinical trial.

Primary Endpoint: total amount of fentanyl consumed during hospital admission. Secondary Endpoints: 1) phase I recovery time; and, 2) time to fitness for discharge.

Exploratory Endpoints: 1) intraoperative hemodynamics; 2) intraoperative opioid use; 3) intraoperative sevoflurane use; 4) postoperative pain; 5) postoperative sedation and cognitive recovery 6) time to first request for analgesia; and, 7) incidence of nausea and vomiting between the end of anesthesia and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older;
* Scheduled for elective knee arthroscopy without anticipated ligamentous repair;
* Planned general anesthesia without a regional block or wound infiltration with local anesthesia;
* Planned day-of-surgery discharge.

Exclusion Criteria:

* Opioid tolerance defined by ≥15 mg of oral morphine daily or equianalgesic dose of another opioid within 30 days of surgery;
* Known hypersensitivity to sufentanil or components of DSUVIA;
* Patients with an allergy or hypersensitivity to opioids;
* Pregnancy or actively breastfeeding;
* Patients who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 14 days of the first dose of study drug;
* Patients with a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including chronic pain or active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabry Ayad, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 35 | 26
Completed | 35 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 35 | 26 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.4) | 51.5 (12.3) | 53.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 20 | 16 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 25 | 60
  non-White | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.9 (5.2) | 33.8 (7.4) | 31.6 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Total Consumption of Fentanyl
Description: The total amount of fentanyl consumed in PACU.
Time Frame: About 3 hours in PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 35 | 26
Participants
  0 µg | 25 | 11
  25 µg | 4 | 5
  50 µg | 2 | 5
  100 µg | 4 | 4
  150 µg | 0 | 1
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.067, proportional odds logistic regression; In the analysis, 100 µg and 150 µg were merged as one level since too few cases used 150 µg; Proportional odds ratio = 0.37, 95% CI 2-sided [0.13 to 1.07]

2. Secondary Outcome: Phase 1 Recovery Time
Description: Recovery will be considered complete at the time an order is placed for progression to phase II.
Time Frame: 1.5 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 35 | 26
minutes | 77 (30) | 66 (18)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.147, Regression, Linear; Mean Difference (Final Values) = 10, 97.5% CI 2-sided [-5.8 to 26]

3. Secondary Outcome: Time to Fitness for PACU Discharge
Description: This will be determined per facility protocol-scheduled assessments using the CCF Phase II Discharge Scoring tool. The time that the minimum acceptable score of 14 is achieved will be recorded
Time Frame: 1 - 2 hours.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 35 | 26
minutes | 120 (47) | 114 (31)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.463, Regression, Linear; Mean Difference (Final Values) = 8.4, 97.5% CI 2-sided [-18 to 34]

4. Other Pre Specified Outcome: Total Consumption of Fentanyl in PACU
Description: The total amount of fentanyl consumed in PACU.
Time Frame: About 3 hours in PACU
Measure: Median (Inter-Quartile Range); unit: µg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 35 | 26
µg | 0 [0 to 25] | 25 [0 to 50]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -13, 95% CI 2-sided [-25 to 0]

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/26
Other Adverse Events (participants affected / at risk) | 0/35 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04561375/Prot_SAP_000.pdf